CLINICAL TRIAL: NCT01573936
Title: The Influence of Rehabilitation on Quality of Life in Adult Patients With Neurological Disorders
Brief Title: Quality of Life in Adult Neurological Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associação de Assistência a Criança Deficiente (Other)
Responsible Party: Principal Investigator, Denise Midori Yoshihara, Principal Investigator, Associação de Assistência a Criança Deficiente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yoshihara_AACD2011
Record Dates: First submitted 2012-03-13; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Spinal Cord Injury; Acquired Brain Injury; Poliomyelitis
Keywords: acquired brain injury; health-related quality of life; poliomyelitis survivor; rehabilitation; spinal cord injury; completed the WHOQOL-BREF
MeSH Terms: conditions — Spinal Cord Injuries; Brain Injuries; Poliomyelitis | interventions — Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rehabilitation program (Experimental): Rehabilitation program from January 2008 through July 2010, which consists of 40-minutes of many therapies for 1-2 days a week
  Interventions: Other: Physical therapy, occupational therapy, psycotherapy, medical consultations

INTERVENTIONS:
Other: Physical therapy, occupational therapy, psycotherapy, medical consultations — The mean duration of the RP was 7.47 ± 4.45 months, but it was not standardized because this factor was not one of the parameters of interest for this study

SUMMARY:
The purposes of this study were to evaluate the influence of an interdisciplinary rehabilitation program in the improvement of the health-related quality of life among adult neurological patients and to identify the sociodemographic and clinical associated characteristics. Subjects with spinal cord injury, acquired brain injury and poliomyelitis survivors participated in the study. All participants underwent a rehabilitation program (RP) from January 2008 through July 2010, which consists of 40-minutes of many therapies for 1-2 days a week. The WHOQOL-BREF was applied at the initial and discharge assessments.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with spinal cord injury, acquired brain injury and poliomyelitis survivors
* at least 18 years old
* consented to participate in the study

Exclusion Criteria:

* cognitive problems to understand and to respond the assessment instrument, according to medical files description and interviewer previous judgment

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF | participants will be followed for the duration of rehabilitation program, an expected average of 7 months
  The brief version of the World Health Organization Quality of Life (WHOQOL-BREF) is a sound, cross-culturally valid assessment of health-related quality of life in adults populations. Its assessment shows good to excellent internal consistency, test-retest reliability, discriminant validity, content validity, and construct validity in the healthy population and in different patient groups.